CLINICAL TRIAL: NCT04764292
Title: Screening Contrast-Enhanced Mammography as an Alternative to MRI
Acronym: SCEMAM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wendie Berg (Other)
Collaborators: PA Breast Cancer Coalition (Unknown)
Responsible Party: Sponsor-Investigator, Wendie Berg, Professor, Department of Radiology, Breast Imaging Division, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY20110029
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: breast cancer supplemental screening; breast density; contrast-enhanced mammography; screening mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Contrast-enhanced mammography (Experimental): Women who meet criteria for supplemental screening MRI, but who are unable to have MRI for medical/access/cost reasons, will be invited to have screening with contrast-enhanced mammography. Women will also have standard-of-care mammography/tomosynthesis per usual clinical practice.
  Interventions: Device: Contrast-enhanced mammography; Drug: Iodinated Contrast Media (ICM)

INTERVENTIONS:
Device: Contrast-enhanced mammography — supplemental breast cancer screening with contrast-enhanced mammography
Drug: Iodinated Contrast Media (ICM) — supplemental breast cancer screening with contrast-enhanced mammography

SUMMARY:
There are women for whom a screening breast MRI is clinically recommended, but not feasible either due to patient factors (body habitus, pacemaker or other implant, claustrophobia) or access (cost, other constraints). Contrast-enhanced mammography (CEM) is a potential alternative to MRI for screening that uses updated standard mammography equipment to obtain low- and high-energy images after intravenous injection of iodinated contrast (as used in CT scanning). The investigators seek to validate screening CEM as an alternative to screening MRI.

DETAILED DESCRIPTION:
This is a prospective study designed to evaluate the role of contrast enhanced mammography (CEM) in screening for breast cancer. The overarching goal of the research program is to improve cancer detection on screening, particularly in women with dense breasts. MRI depicts more cancers than other screening methods, including ultrasound. MRI is proven to both improve cancer detection and reduce clinically detected cancers ("interval cancers") after a negative screening mammogram in women with dense breasts. PA Senate Bill 595, signed into law June 30, 2020, requires insurance carriers to provide coverage for supplemental screening with MRI or ultrasound for a variety of indications. Relative to the number of women who may benefit from screening MRI, there is a shortage of equipment/capacity. Further, nearly half of women cannot have an MRI for medical or other reasons, such as claustrophobia, implanted devices, body habitus, or cost (deductible and copay apply even with the new legislation). Contrast-enhanced mammography (CEM) appears to have similar performance to MRI but has not been widely validated, particularly for screening. In order to lay the foundation for improved screening of women with dense breasts, the investigators seek to offer screening CEM as an alternative to MRI for women who meet guidelines for screening MRI but are unable to have MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic women under age 75 who are recommended for annual screening MRI and mammography based on current criteria:

   1. Women known to be at high risk for breast cancer because of known or suspected pathogenic mutation, prior chest radiation therapy at least 8 years earlier and before age 30, or estimated lifetime risk of at least 20% based on family history/prior biopsy history (22), between age 30 and 75.
   2. Women with extremely dense breasts age 40-75 (about 7% of the screening population (1)) (12).
2. Women with lobular carcinoma in situ (1% of women biopsied each year; about 0.06% of our screening population) beginning the year after diagnosis.
3. Women with a personal history of breast cancer diagnosed by age 50 or with dense breasts (21), beginning the year after diagnosis (will be recruited under separate ongoing TOCEM protocol).
4. Women with heterogeneously dense breasts and any family history of breast cancer (about 36% of the screening population has dense breasts and about 20% have a family history of breast cancer) who do not meet current high-risk criteria, beginning at age 40 or ten years prior to the age of the youngest relative but not before age 30.

Participants are expected to have medical or other reasons that they are not able to have screening breast MRI.

Exclusion Criteria:

1. Under age 30 or over age 75.
2. Pregnant or breast feeding.
3. Breast implants.
4. Breast surgery within the prior 12 months.
5. Breast signs or symptoms (lump, nipple discharge, nipple retraction, or being followed for breast abnormality on prior imaging).
6. Currently undergoing any type of systemic chemotherapy for cancer (excludes oral endocrine therapy such as aromatase inhibitors or tamoxifen).
7. Reduced kidney function with eGFR < 45 mL/min.

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Cancer Detection Rate | 1.5 years
  To show significantly improved cancer detection with CEM compared to standard mammography/tomosynthesis

SECONDARY OUTCOMES:
False Positive Recall Rates | 1.5 years
  To show acceptably low false positive recall rates from CEM.

CONTACTS AND LOCATIONS:
Overall Officials: Wendie Berg, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - UPMC Magee at the Lemieux Sports Complex, Cranberry Township, Pennsylvania
  - UPMC Magee Monroeville Breast Care Center, Pittsburgh, Pennsylvania
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Images may be shared with secondary investigators, including commercial companies after removal of all identifiers. All patient identification (name, patient number, birth date) will be removed from the DICOM headers of the images.
Time Frame: after publication
Access Criteria: secondary investigators for image analysis. Sharing via Box

REFERENCES:
- [Derived] Berg WA, Vargo A, Lu AH, Berg JM, Bandos AI, Hartman JY, Zuley ML, Ganott MA, Kelly AE, Nair BE, Chough DM, Reginella RF, Wallace LP, Harnist KS, Carlin BA, Cohen CS, Hakim CM, Sumkin JH. Screening for Breast Cancer with Contrast-enhanced Mammography as an Alternative to MRI: SCEMAM Trial Results. Radiology. 2025 Jun;315(3):e242634. doi: 10.1148/radiol.242634. PMID 40525975